CLINICAL TRIAL: NCT06351436
Title: Using Mindfulness With Immersive Virtual Reality Cave Experience in Promoting Mental Well-Being: A Feasibility Study
Brief Title: Virtual Reality Cave Experience With Mindfulness for Mental Wellbeing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TBC20240402
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Anxiety
Keywords: Anxiety; Mental Well-Being; Mindfulness-Based Intervention; Virtual Reality; Youths
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Single-group non-randomized uncontrolled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — The mindfulness-based intervention will last for three months, with 6-8 weekly sessions lasting 1.5 hours each. Participants will attend the sessions in a group format, and the sessions will be administered by registered social worker who are specialized in counseling. The intervention is delivered using an immersive virtual reality cave system. The intervention content is designed by a registered clinical psychologist accredited for delivering mindfulness-based intervention and nurses who are experienced in mindfulness training. To ensure protocol adherence, the social workers administering the intervention will receive close supervision from the clinical psychologist. Weekly meetings will be held to discuss and resolve any difficulties or challenges encountered by the social workers.

SUMMARY:
The aim of this study is to investigate the effectiveness of a mindfulness-based intervention using a virtual reality cave system for promoting mental wellbeing in youths. The mindfulness-based intervention will last for three months, with 6-8 weekly sessions lasting 1.5 hours each. Participants will attend the sessions in a group format, and the sessions will be administered by registered social worker who are specialized in counselling. The intervention content is designed by a registered clinical psychologist accredited for delivering mindfulness-based intervention and nurses who are experienced in mindfulness training.

A single-group pre-post uncontrolled design will be employed. Evaluations will be conducted at baseline (0 weeks) and post-intervention (3 months).

DETAILED DESCRIPTION:
Anxiety disorders in youths are associated with poorer social relationships and academic achievements. If left unaddressed, youth anxiety disorders can progress into adult anxiety disorders, depression, substance abuse, suicide attempts, and hospitalization. Mindfulness-based interventions show promise as an intervention for targeting anxiety symptoms in youths. Recently, virtual reality has emerged as an appealing modality for delivering mindfulness-based interventions. Compared to traditional delivery methods, virtual reality offers a highly engaging and interactive environment for mindfulness practice, allowing users to fully immerse themselves in the virtual setting and minimizing distractions from the physical world. As an innovative pedagogical tool, virtual reality provides an experiential learning environment for mindfulness training, facilitating the cultivation of mindfulness skills through immersive experiences. Preliminary evidence suggests that virtual reality-based mindfulness-based interventions can effectively reduce anxiety symptoms in clinical populations. However, it remains unclear whether these findings can be generalized to a younger population. This pilot feasibility study aims to investigate the effectiveness of a virtual reality-based mindfulness-based intervention in reducing anxiety symptoms among this specific population.

A single-group pre-post uncontrolled design will be employed. The target population for this study will be Hong Kong Chinese youths with mild to moderate anxiety symptoms. Convenience sampling will be used to recruit participants. Interested participants will be assessed for eligibility. After interested and eligible participants provide their consent, they will receive the mindfulness-based intervention using a virtual reality cave system.

The mindfulness-based intervention will last for three months, with 6-8 weekly sessions lasting 1.5 hours each. Participants will attend the sessions in a group format, and the sessions will be administered by registered social worker who are specialized in counselling. The intervention is delivered using an immersive virtual reality cave system. The intervention content is designed by a registered clinical psychologist accredited for delivering mindfulness-based intervention and nurses who are experienced in mindfulness training. To ensure protocol adherence, the social workers administering the intervention will receive close supervision from the clinical psychologist. Weekly meetings will be held to discuss and resolve any difficulties or challenges encountered by the social workers.

The outcome measures assessed included mental wellbeing (primary) and heart rate variability (secondary). Feasibility measures include eligibility and enrollment, attendance rate, and retention rate. Evaluations will be conducted at baseline (0 weeks) and post-intervention (3 months).

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese youths;
* aged between 11 and 18;
* screened positive for mild to moderate anxiety symptoms (a summed score of ≥ 10 as measured by the Generalized Anxiety Disorder-7).

Exclusion Criteria:

* screened positive for clinical depression (a summed score of ≥ 9 as measured by the Patient Health Questionnaire-9).

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Mental Well-Being in Youths | 3 months
  The Depression Anxiety Stress Scale-21 (DASS) consists of 21 items that assess three domains: anxiety, depression, and stress. Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all) to 3 (applied to me much or most of the time). The total score for each subscale ranges from 0 to 21, with higher scores indicating greater severity in the respective domain.

SECONDARY OUTCOMES:
Stress Level in Youths | 3 months
  Heart rate variability is a measure of the variation in the time intervals between consecutive heartbeats and is commonly used as an indicator of stress levels. To assess heart rate variability, we utilized Upmood®, a wearable device equipped with a photoplethysmogram (PPG) sensor. This device enables non-invasive measurement of HRV by analyzing pulse signal power and calculating various indices such as HF (high frequency), LF (low frequency), LF/HF ratio, and VLF (very low frequency), with a lower level of heart rate variability indicating a higher level of stress.
Feasibility of Eligibility and Enrollment | 3 months
  Number of eligible participants, and the proportion of those eligible that enrolled will be assessed.
Feasibility of Attendance Rate | 3 months
  Number and proportion of attended participants.
Feasibility of Retention Rate | 3 months
  Number and proportion of participants completing all assessments.

IPD SHARING:
Plan to Share IPD: No